CLINICAL TRIAL: NCT07074236
Title: A Randomized, Open-label, Single-center, Parallel Study in Subjects With Normal or Elevated Low-density Lipoprotein Cholesterol Level to Compare the Pharmacokinetics and Pharmacodynamics of the Two Formulations of QLC7401 Injection
Brief Title: Pharmacokinetics and Pharmacodynamics Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLC7401-102
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Primary Hypercholesterolemia or Combined Hyperlipidemia Characterized by Elevated LDL-C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLC7401 injection (Experimental)
  Interventions: Drug: QLC7401 injection
- RBD7022 injection (Experimental)
  Interventions: Drug: RBD7022 injection

INTERVENTIONS:
Drug: QLC7401 injection — QLC7401 injection is a small interfering RNA (siRNA) directed to PCSK9 (proprotein convertase subtilisin kexin type 9) mRNA to inhibit the translation of PCSK9 and reduce expression of PCSK9 protein further to lower the level of LDL-C. QLC7401 injection was introduced by Qilu Pharmaceutical Co., Ltd. from Suzhou Ruibo Biotechnology Co., Ltd. QLC7401 injection was produced by Qilu Pharmaceutical Co., Ltd.
  Arms: QLC7401 injection
Drug: RBD7022 injection — RBD7022 injection is a small interfering RNA (siRNA) directed to PCSK9 (proprotein convertase subtilisin kexin type 9) mRNA to inhibit the translation of PCSK9 and reduce expression of PCSK9 protein further to lower the level of LDL-C. RBD7022 injection was produced by Suzhou Ruibo Biotechnology Co., Ltd.
  Arms: RBD7022 injection

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and pharmacodynamics behavior of the two formulation of QLC7401 injection to further evaluate the effect of the production site change.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are 18 to 65 years of age.
* BMI is within the range of 18~28 kg/m2 (including the boundary value).
* LDL-C is within the range of 1.8 mmol/L (70 mg/dl) and 4.1 mmol/L (158 mg/dl) (including the lower boundary value). TG is less than or equal to 4.5 mmol/L (400 mg/dl).
* TC is less than 6.2 mmol/L (239 mg/dl).

Exclusion Criteria:

* Subjects with confirmed diabetes.
* Subjects with severe active psychiatric illness or disorder.
* eGFR is less than 90 ml/min.
* AST is equal to or above the 2 fold of upper limit of normal value or TBIL is equal to or above the 1.5 fold of upper limit of normal value.
* Subjects administered prescription drugs 14 days before the first drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Maximum plasma concentration of QLC7401 and active metabolites.
AUC | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Area under the concentration-time curve of QLC7401 and active metabolites.
Tmax | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Time of maximum observed concentration of QLC7401 and active metabolites..
t1/2 | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Terminal elimination half-life of QLC7401 and active metabolites.
CL/F | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Apparent total clearance of the drug from plasma after oral administration of QLC7401 and active metabolites.
VZ/F | 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post dose
  Apparent volume of distribution after oral administration of QLC7401 and active metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University., Qingdao, China